CLINICAL TRIAL: NCT02422654
Title: A Single-blind, Randomized, Unbalanced Crossover Design With 5 Vehicles, 5 Periods, and 5 Sequences, Repeated-doses (With no Ingestion) Study to Assess the Palatability of Eliglustat Prototype Liquid Formulations in Healthy Subjects
Brief Title: Taste Evaluation of Different Liquid Formulations With Eliglustat
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: ACC14373; U1111-1168-5133 (Other: UTN)
Record Dates: First submitted 2015-04-14; First posted 2015-04-21 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Gaucher Disease
MeSH Terms: conditions — Gaucher Disease | interventions — eliglustat

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (15):
- Concentration 1 eliglustat in vehicle A (Experimental): Single dose of 5 mL solution held in the mouth for 15 seconds with swishing but with no ingestion
  Interventions: Drug: eliglustat
- Concentration 1 eliglustat in vehicle B (Experimental): Single dose of 5 mL solution held in the mouth for 15 seconds with swishing but with no ingestion
  Interventions: Drug: eliglustat
- Concentration 1 eliglustat in vehicle C (Experimental): Single dose of 5 mL solution held in the mouth for 15 seconds with swishing but with no ingestion
  Interventions: Drug: eliglustat
- Concentration 1 eliglustat in vehicle D (Experimental): Single dose of 5 mL solution held in the mouth for 15 seconds with swishing but with no ingestion
  Interventions: Drug: eliglustat
- Concentration 1 eliglustat in vehicle E (Experimental): Single dose of 5 mL solution held in the mouth for 15 seconds with swishing but with no ingestion
  Interventions: Drug: eliglustat
- Concentration 2 eliglustat in vehicle A (Experimental): Single dose of 5 mL liquid formulation held in the mouth for 15 seconds with swishing but with no ingestion
  Interventions: Drug: eliglustat
- Concentration 2 eliglustat in vehicle B (Experimental): Single dose of 5 mL liquid formulation held in the mouth for 15 seconds with swishing but with no ingestion
  Interventions: Drug: eliglustat
- Concentration 2 eliglustat in vehicle C (Experimental): Single dose of 5 mL liquid formulation held in the mouth for 15 seconds with swishing but with no ingestion
  Interventions: Drug: eliglustat
- Concentration 2 eliglustat in vehicle D (Experimental): Single dose of 5 mL liquid formulation held in the mouth for 15 seconds with swishing but with no ingestion
  Interventions: Drug: eliglustat
- Concentration 2 eliglustat in vehicle E (Experimental): Single dose of 5 mL liquid formulation held in the mouth for 15 seconds with swishing but with no ingestion
  Interventions: Drug: eliglustat
- Concentration 3 eliglustat in vehicle A (Experimental): Single dose of 5 mL liquid formulation held in the mouth for 15 seconds with swishing but with no ingestion
  Interventions: Drug: eliglustat
- Concentration 3 eliglustat in vehicle B (Experimental): Single dose of 5 mL liquid formulation held in the mouth for 15 seconds with swishing but with no ingestion
  Interventions: Drug: eliglustat
- Concentration 3 eliglustat in vehicle C (Experimental): Single dose of 5 mL liquid formulation held in the mouth for 15 seconds with swishing but with no ingestion
  Interventions: Drug: eliglustat
- Concentration 3 eliglustat in vehicle D (Experimental): Single dose of 5 mL liquid formulation held in the mouth for 15 seconds with swishing but with no ingestion
  Interventions: Drug: eliglustat
- Concentration 3 eliglustat in vehicle E (Experimental): Single dose of 5 mL liquid formulation held in the mouth for 15 seconds with swishing but with no ingestion
  Interventions: Drug: eliglustat

INTERVENTIONS:
Drug: eliglustat — Pharmaceutical form:liquid formulation
  Route of administration: oral without ingestion
  Other Names: GZ385660

SUMMARY:
Primary Objective:

The purpose of this study is to assess the palatability of eliglustat prototype liquid formulations in healthy subjects.

DETAILED DESCRIPTION:
The total duration of the study for each subject will be approximately 5 weeks (screening period from Day -28 to Day -2, treatment period of 3 days, and follow-up call on Day 5).

ELIGIBILITY:
Inclusion criteria :

* Healthy male and female subjects, 18 to 55 years of age, inclusive.
* Normal smell and taste ability to discriminate odor and flavor differences.

Exclusion criteria:

* Poor metabolizer phenotype status for CYP2D6 (predicted based on genotype).
* Subject who has smoked within 3 months of inclusion.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2015-04; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Measurement of palatability by 100 mm visual analogue scale (VAS) for overall acceptability | Each day for 3 days immediately post expectorating the sample
Measurement of palatability by 100 mm visual analogue scale (VAS) for overall acceptability | Each day for 3 days 5 minutes post expectorating the sample
Measurement of palatability by 100 mm visual analogue scale (VAS) for overall acceptability | Each day for 3 days 15 minutes post expectorating the sample
Measurement of palatability by 100 mm visual analogue scale (VAS) for overall acceptability | Each day for 3 days 30 minutes post expectorating the sample

SECONDARY OUTCOMES:
Subject's taste preference questionnaire from most preferred to least preferred of the 5 different liquid formulations | up to 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site Number 840001, Evansville, Indiana, United States